CLINICAL TRIAL: NCT00843050
Title: Single-Arm, Open-Label, Multicenter Phase II Study to Evaluate the Efficacy and Safety of P276-00 in Patients With Relapsed and/or Refractory Mantle Cell Lymphoma
Brief Title: A Phase II Study to Evaluate Efficacy and Safety of P276-00 in Relapsed and/or Refractory Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on interim results and all subjects were off study at that time. No major safety or tolerability concerns
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/23/08
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: CKD inhibitor; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- P276-00 (Experimental): P276-00: All patients will receive P276-00 185 mg/m2/day as intravenous infusion over 30 minutes in 200 ml of 5% dextrose from day 1 to day 5 in each 21 days cycle for minimum 6 and maximum 12 cycles or until there is progression of disease or unacceptable toxicity
  Interventions: Drug: P276-00

INTERVENTIONS:
Drug: P276-00 — P276-00: All patients will receive P276-00 185 mg/m2/day as intravenous infusion over 30 minutes in 200 ml of 5% dextrose from day 1 to day 5 in each 21 days cycle for minimum 6 and maximum 12 cycles or until there is progression of disease or unacceptable toxicity

SUMMARY:
The purpose of this study is to determine whether P276-00 is safe and effective in treatment of Mantle Cell Lymphoma that is recurred after or not responding to at least one previous line of treatment.

DETAILED DESCRIPTION:
Despite response rates of up to 97% with first-line standard or high-intensity chemotherapy, with or without stem-cell transplantation, most patients of mantle cell lymphoma (MCL)relapse.Prognosis of MCL after first relapse is very poor with median survival of around 1 to 2 years. Therefore, novel therapies are required for relapsed and/or refractory MCL.Overexpression of Cyclin D1 as a result of t(11;14)(q13;q32) translocation is the hallmark of MCL.It is postulated that Cyclin D1 may also have an oncogenic role independent of pRb in MCL.Therefore, inhibition of Cdk4-Cyclin D1 is a potentially promising target in MCL. P276-00 is a potent Cdk4-Cyclin D1 inhibitor worth exploring for its efficacy in MCL. Hence, this Phase II study is planned to examine the efficacy and safety of P276-00 in the treatment of patients with relapsed and/or refractory MCL.

This is an open-label, single-arm, 2-stage trial. Approximately 35 patients are planned to be enrolled into the study to obtain a total of 25 efficacy evaluable patients (patients who complete at least 2 cycles of study treatment and have tumor measurements at the end of 2 cycles). A total of 15 efficacy evaluable patients are planned to be treated in Stage I of the study. If ≥1 response (CR or PR) of any duration or ≥2 stable disease (SD) for ≥4 cycles are seen in the Stage I, then the study will continue into Stage II, in which additional patients will be treated until there are 10 additional efficacy evaluable patients.The study is divided into 3 periods: Screening, Treatment, and Follow-up. During the Screening Period, patients will provide written informed consent and be evaluated for inclusion and exclusion criteria. During the Treatment Period, patients will be administered P276-00 as intravenous (iv) infusion on Days 1 to 5 of each 21-day cycle for a minimum of 6 cycles and a maximum of 12 cycles, or until progressive disease (PD) or unacceptable toxicity occurs. Safety and efficacy evaluations will be done on Days 1 to 5 and 11 of each cycle, and on Day 21 of every 2 cycles. Pharmacokinetic (PK) assessments will be done on Cycle 1, Day 1 (pre-dose and post-dose time points), and optional biomarker assessments will be done pre-dose within 4 weeks of Day 1 and post-dose on Day 4 or 5. The End-of-Last-Cycle Visit will occur at the end of Cycle 6, or if the patient continues study treatment beyond Cycle 6, it will occur at the end of the patient's last cycle; if the patient discontinues early, these assessments will be done as an Early Exit Visit. The Follow-up Visit will occur 4 weeks (±1 week) after the End-of-Last-Cycle Visit (or Early Exit Visit) for final safety assessments.Objective response rate is the primary end point for this study. Response evaluation will be performed using the International Working Group (IWG) revised response criteria for malignant lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histological diagnosis of MCL and presence of either nuclear Cyclin D1 positivity by immunohistochemistry or t(11;14) by fluorescence in situ hybridization (FISH), polymerase chain reaction (PCR), or conventional karyotyping
* Documented progression or relapse after at least 1 line of prior chemotherapy
* Presence of measurable disease
* ECOG performance status 0, 1, or 2
* Life expectancy of at least 3 months
* Ability to understand and the willingness to sign a written informed consent document (ICD)
* Full recovery from all prior treatment toxicities of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1

Exclusion Criteria:

* Prior radiation therapy, chemotherapy or biologic/targeted anticancer agents within 4 weeks of study drug administration
* Prior treatment with monoclonal antibodies or any radio- or toxin- immunoconjugates within 3 months of study drug administration; however, a patient who has had rituximab treatment within 3 months and has had PD after such treatment is allowed in the study.
* Prior allogeneic stem cell transplantation within 1 year of study drug administration
* Current or prior CNS lymphoma
* QTc > 450 msec
* Unstable angina, myocardial infarction, CHF or stroke within previous 6 months of study drug administration
* Presence of active and serious comorbidity and uncontrolled illness other than MCL
* History of other prior malignancies except for properly treated basal cell or squamous cell carcinoma of skin, in situ cervical cancer, in situ breast cancer or early stage prostate cancer
* Hemoglobin <8.0 gm/dL
* Absolute neutrophil count <1000/mm3
* Platelet count <50,000/mm3
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >3 × institutional upper limit of normal (ULN) (> 5 × institutional ULN if liver is involved with lymphoma or if patient has Gilbert's Disease)
* Total bilirubin, >1.5 × institutional ULN (> 3 × institutional ULN if liver is involved with lymphoma or if patient has Gilbert's Disease)
* Serum creatinine >1.5 × institutional ULN
* Patients known to be suffering from infection with human immunodeficiency virus (HIV), tuberculosis, Hepatitis C or Hepatitis B
* Pregnant or lactating women
* Women of childbearing potential or men not willing to use at least 2 approved methods of contraception (one of which being a barrier method) after signing the ICD, during the entire study and for at least 4 weeks following withdrawal from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Kahl, MD, Principal Investigator — Director of the Lymphoma Service and Associate Professor of Medicine, University of Wisconsin- Madison; Gabrail Nashat, MD, Principal Investigator — CEO, President, Gabrail Cancer Center; Martha Glenn, MD, Principal Investigator — Associate Professor of Medicine, Huntsman Cancer Institute, Salt Lake City; Andre Goy, MD, Principal Investigator — Director of Lymphoma and Deputy Director of Cancer Center, Hackensack University Medical Center, Hackensack; Roger Lyons, MD, Principal Investigator — President, Cancer Care Centers of South Texas , San Antonio; Nishitha Reddy, MD, Principal Investigator — Vanderbilt University Medical Center, Nashville; Reena Nair, MD, Principal Investigator — Professor and Medical Oncologist, Tata Memorial Hospital, Mumbai, India; Anand Pathak, MD, Principal Investigator — Medical Oncologist, Cancer Care Clinic and Hospital, Nagpur, India; Vinod Raina, MD, Principal Investigator — Head Dept of Medical Oncology, Institute Rotary Cancer Hospital, All India Institute of Medical Sciences, New Delhi, India; N K Warrier, MD, Principal Investigator — Senior Consultant Oncologist, Malabar Institute of Medical Sciences, Calicut, India; Cecil Ross, MD, Principal Investigator — Consultant Oncologist, St. Johns Medical College & Hospital, Bangalore, India; Kirushna kumar, MD, Principal Investigator — Consultant Oncologist, Meenakshi mission hospital and research centre, Madurai, India; S H Advani, MD, Principal Investigator — Consultant Oncologist, Jaslok Hospital and Research Centre, Mumbai, India; Patrick Johnston, MD, Principal Investigator — Associate Professor of Medicine, College of Medicine, Mayo Clinic, Rochester, USA; Ajay Gopal, MD, Principal Investigator — Associate Professor of Medicine, Department of Medicine, University of Washington, Seattle, Washington.; Craig Reeder, MD, Principal Investigator — Consultant, Division of Hematology/Oncology, Department of Internal Medicine, Mayo Clinic, Arizona
Locations (20):
- United States (13):
  - Division of Hematology/Oncology, Department of Internal Medicine, Mayo Clinic, Phoenix, Arizona, Phoenix, Arizona
  - Division of Hematology/Oncology, Department of Internal Medicine, Mayo Clinic, Arizona, Scottsdale, Arizona
  - College of Medicine, Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Gabrail Cancer Center Research, Canton, Ohio
  - Gabrail Cancer Center Research, Dover, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cancer Care Centers of South Texas, New Braunfels, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Huntsman Cancer Institute, 2000 Circle of Hope, Room 2145, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Department of Medicine, University of Washington, Seattle, Washington
  - Dept of Hematology/Oncology, University of Wisconsin- Madison, Madison, Wisconsin
- India (7):
  - St. Johns Medical College & Hospital, Bangalore, Karnataka
  - Malabar Institute of Medical Sciences, Calicut, Kerala
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Cancer Care Clinic and Hospital, Nagpur, Maharashtra
  - Institute Rotary Cancer Hospital, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Meenakshi mission hospital and research centre, Madurai, Tamil Nadu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across multiple centers in the United States and India.
Period: Overall Study
Arm/Group | P276-00
Started | 13
Completed | 0
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | P276-00
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 65.8 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 8
  India | 5

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Objective Response Rate
Description: The primary efficacy endpoint is the proportion of subjects achieving an objective response. The proportion of patients achieving an objective response is the best overall objective response rate.
Time Frame: End of every 2 cycles and end of the study treatment
Population: The efficacy population includes all patients who have completed at least two cycles of P276-00 therapy and have tumor measurements.
Measure: Mean (Standard Deviation); unit: proportion of participants
Groups:
- P276-00: P276-00: All patients received P276-00 185 mg/m2/day as intravenous infusion over 30 minutes in 200 ml of 5% dextrose from day 1 to day 5 in each 21 days cycle for minimum 6 and maximum 12 cycles or until there was progression of disease or unacceptable toxicity
Arm/Group | P276-00
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Description: It is defined as the time from when the measurement criteria are met for complete or partial response until the first date that recurrent or progressive disease is objectively or clinically documented.
Time Frame: End of the study treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Arm/Group | P276-00
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Progression
Description: It is defined as the time from day 1 of the study drug administration until the first date of progressive disease.
Time Frame: End of study treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: years
Arm/Group | P276-00
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | P276-00
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P276-00 (N=13)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Disease Progression (General disorders) | 2 (2)
Elevated Creatinine, (Renal and urinary disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P276-00 (N=13)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Arthropod bite (Infections and infestations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Asthenia (General disorders) | 1 (1)
Blood Alkaline Phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Cardiac murmur (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Decrreased Appetite (Gastrointestinal disorders) | 2 (2)
Dehydration (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (6)
Dizziness (Nervous system disorders) | 2 (2)
Dry Eye (Eye disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Electrocardiogram QT prolonged (Cardiac disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 4 (5)
Gastritis (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 6 (10)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
Injection site swelling (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2)
Lymphadenopathy (General disorders) | 1 (1)
Left atrial dilatation (Cardiac disorders) | 1 (1)
lymphocyte count increased (Investigations) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (7)
nausea (Gastrointestinal disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (2)
neutrophil count decreased (Investigations) | 1 (1)
nocturia (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema (General disorders) | 2 (4)
Oedema peripheral (General disorders) | 5 (5)
pain (General disorders) | 1 (1)
Pain in extremity (General disorders) | 2 (2)
Panic attack (Nervous system disorders) | 1 (1)
Penile swelling (General disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pollakiuria (Metabolism and nutrition disorders) | 1 (1)
Post operative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Pruritus (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Rash Pruritic (General disorders) | 1 (1)
Rash pustular (General disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2)
skin burning sensation (General disorders) | 1 (1)
spleen palpable (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor has terminated the study based on interim results. All subjects were off study at the time of termination. There are no major safety or tolerability concerns from this study. The study results published here are preliminary results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No